CLINICAL TRIAL: NCT03043274
Title: Periprocedural Cangrelor in Patients With ST-Elevation Myocardial Infarction to Reduce Development of Myocardial Necrosis
Brief Title: Cangrelor in ST-Elevation Myocardial Infarction to Decrease Infarct Size
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Khaled Ziada, MD (Other)
Responsible Party: Sponsor-Investigator, Khaled Ziada, MD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0990-F6A
Record Dates: First submitted 2017-01-15; First posted 2017-02-06 (Estimated); Results first posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — cangrelor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cangrelor (Experimental): Approximately 30 patients in this arm will receive standard STEMI care but will also receive standard dosing of cangrelor at the time of their PCI.
  Interventions: Drug: Cangrelor
- No cangrelor (No Intervention): Approximately 30 patients in this arm will receive standard STEMI but will not receive cangrelor at the time of their PCI.

INTERVENTIONS:
Drug: Cangrelor — Cangrelor 30 mcg/kg bolus followed by a 4 mcg/kg/min intravenous infusion prior to PCI will be given. It will be continued for ≥ 2 hours or for the duration of the procedure, whichever is longer.
  Other Names: Kengreal
  Arms: Cangrelor

SUMMARY:
This study evaluates differences in the extent of myocardial necrosis noted by cardiac MRI in patients with ST-elevation myocardial infarction randomized to receive cangrelor during their percutaneous coronary intervention and compares them to patients randomized to not receive cangrelor.

DETAILED DESCRIPTION:
Cangrelor is a direct-acting and reversible intravenously administered platelet inhibitor approved as an adjunct to percutaneous intervention (PCI) for reducing the risk of periprocedural myocardial infarction, repeat coronary revascularization, and stent thrombosis. As it has a quick onset of action (2 minutes) compared to traditional oral platelet inhibitors, cangrelor is emerging as an important new option for use in patients undergoing percutaneous intervention who have not been treated with oral platelet inhibitors.

Furthermore, multiple studies have demonstrated that patients with ST-elevation myocardial infarction (STEMI) who undergo emergent PCI do not have optimal platelet inhibition even after administration of a loading dose of traditional oral platelet inhibitors. However, the clinical significance of complete platelet inhibition around the time of PCI is not fully understood.

The primary objective is to characterize the utility of immediate platelet inhibition with intravenous cangrelor in patients presenting with an acute STEMI by assessing the extent of infarct size (either enzymatically or by imaging). If the findings are favorable, this may suggest that immediate platelet inhibition is an important part of care in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an acute STEMI with the University of Kentucky as the institution of presentation with plans for PCI
* English-speaking

Exclusion Criteria:

* Pregnant patients
* Prisoners
* Patients who are unable to provide his/her own consent
* Patients with a prior history of myocardial infarction
* Patients who have received thrombolytics
* Patients on systemic anticoagulation
* Patients who are hemodynamically unstable with evidence of shock
* Patients who are mechanically intubated
* Patients with devices not MRI compatible
* Patients with chronic kidney disease, glomerular filtration rate less than 30
* Patients who are already on dual antiplatelet therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Ziada, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keating GM. Cangrelor: A Review in Percutaneous Coronary Intervention. Drugs. 2015 Aug;75(12):1425-34. doi: 10.1007/s40265-015-0445-3. PMID 26201463
- [Background] Johnson TW, Mumford AD, Scott LJ, Mundell S, Butler M, Strange JW, Rogers CA, Reeves BC, Baumbach A. A Study of Platelet Inhibition, Using a 'Point of Care' Platelet Function Test, following Primary Percutaneous Coronary Intervention for ST-Elevation Myocardial Infarction [PINPOINT-PPCI]. PLoS One. 2015 Dec 16;10(12):e0144984. doi: 10.1371/journal.pone.0144984. eCollection 2015. PMID 26672598
- [Background] Parodi G, Valenti R, Bellandi B, Migliorini A, Marcucci R, Comito V, Carrabba N, Santini A, Gensini GF, Abbate R, Antoniucci D. Comparison of prasugrel and ticagrelor loading doses in ST-segment elevation myocardial infarction patients: RAPID (Rapid Activity of Platelet Inhibitor Drugs) primary PCI study. J Am Coll Cardiol. 2013 Apr 16;61(15):1601-6. doi: 10.1016/j.jacc.2013.01.024. Epub 2013 Mar 22. PMID 23500251
- [Background] Sibbing D, Braun S, Morath T, Mehilli J, Vogt W, Schomig A, Kastrati A, von Beckerath N. Platelet reactivity after clopidogrel treatment assessed with point-of-care analysis and early drug-eluting stent thrombosis. J Am Coll Cardiol. 2009 Mar 10;53(10):849-56. doi: 10.1016/j.jacc.2008.11.030. PMID 19264241
- [Background] Stone GW, Maehara A, Witzenbichler B, Godlewski J, Parise H, Dambrink JH, Ochala A, Carlton TW, Cristea E, Wolff SD, Brener SJ, Chowdhary S, El-Omar M, Neunteufl T, Metzger DC, Karwoski T, Dizon JM, Mehran R, Gibson CM; INFUSE-AMI Investigators. Intracoronary abciximab and aspiration thrombectomy in patients with large anterior myocardial infarction: the INFUSE-AMI randomized trial. JAMA. 2012 May 2;307(17):1817-26. doi: 10.1001/jama.2012.421. Epub 2012 Mar 25. PMID 22447888
- [Derived] Abo-Aly M, George B, Shokri E, Chelvarajan L, El-Helw M, Smyth SS, Abdel-Latif A, Ziada K. Cangrelor in addition to standard therapy reduces cardiac damage and inflammatory markers in patients with ST-segment elevation myocardial infarction. J Thromb Thrombolysis. 2021 Oct;52(3):934-940. doi: 10.1007/s11239-020-02345-8. Epub 2020 Nov 30. PMID 33258102
- See also: Related Info — http://www.kengreal.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the cardiac catheterization laboratory.
Pre-assignment Details: Patients were randomized upon recruitment to the standard of care alone or standard of care in addition to cangrelor
Groups:
- Cangrelor: Patients received standard of care in addition to cangrelor with a dose of 30 mcg/kg bolus followed by a 4 mcg/kg/min intravenous infusion, started prior to PPCI, and continued for 2 hours or for the duration of the procedure, whichever is longer.
- No Cangrelor: This arm received standard of care alone
Period: Overall Study
Arm/Group | Cangrelor | No Cangrelor
Started | 13 | 10
Completed | 13 (The study was terminated because of slow recruitment.) | 9 (The study was terminated because of slow recruitment.)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cangrelor: The final subject count in this arm is 13.
- No Cangrelor: The final subject number in this arm is 9.
- Total: Total of all reporting groups
Arm/Group | Cangrelor | No Cangrelor | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.7) | 57.4 (7.7) | 58.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.8 (2) | 31.6 (8.1) | 29.96 (7.24)
Diabetes [Count of Participants; unit: Participants] | 3 | 4 | 7
Hypertension [Count of Participants; unit: Participants] | 8 | 6 | 14
Hyperlipidemia [Count of Participants; unit: Participants] | 3 | 4 | 7
Peripehral vascular disease [Count of Participants; unit: Participants] | 2 | 0 | 2
No prior platelet therapy [Count of Participants; unit: Participants] | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Myocardial Infarction Size
Description: Cardiac MRI is obtained at 48 hours and 3 months to compare differences in infarct size. The outcome is assessed as the difference in infarct size between 48 hours and 3 months in each group.
Time Frame: 48 hours and 3 months
Population: standard of care alone vs. Standard of care in addition to cangrelor
Measure: Mean (Standard Error); unit: percent of left ventricular mass
Arm/Group | Cangrelor | No Cangrelor
Number analyzed (Participants) | 13 | 9
percent of left ventricular mass
  48 hours | 8.6 (1.6) | 11.1 (2.1)
  3 months | 6.7 (1.5) | 6.98 (2.1)

2. Secondary Outcome: Platelet Reactivity
Description: Platelet reactivity testing will be performed 10 minutes after infusion has started.
Time Frame: 10 minutes
Population: standard of care alone vs. Standard of care in addition to cangrelor
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Cangrelor | No Cangrelor
Number analyzed (Participants) | 13 | 9
seconds
  ADP-induced aggregation | 102.2 (24.88) | 333.4 (63.3)
  TRAP-induced aggregation | 285.8 (86.1) | 624.8 (106)

3. Secondary Outcome: Peripheral Blood Count Quantification
Description: Flow cytometry on peripheral blood will be performed to quantify peripheral counts of inflammatory cells, stem cells, and monocyte subtypes.
Time Frame: 6 hours
Population: standard of care alone vs. Standard of care in addition to cangrelor
Measure: Mean (Standard Error); unit: cells per microliter
Arm/Group | Cangrelor | No Cangrelor
Number analyzed (Participants) | 13 | 9
cells per microliter
  granulocyte platelet aggregates | 1166.7 (190.7) | 2550.4 (533.7)
  Monocyte-platelet aggregate | 139.8 (31.1) | 333.9 (44.9)

4. Secondary Outcome: Interferon (IFN)-α2
Description: ELISA assay will be performed on plasma to quantify the amount of the inflammatory cytokine interleukin-6 in pg/mL.
Time Frame: 6 hours
Population: Plasma level
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Cangrelor | No Cangrelor
Number analyzed (Participants) | 13 | 9
pg/mL | 33.2 (5.9) | 57.8 (4.6)

5. Secondary Outcome: IFN-γ
Description: ELISA assay.
Time Frame: 6 hours
Population: Plasma levels
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Cangrelor | No Cangrelor
Number analyzed (Participants) | 13 | 9
pg/mL | 41.4 (8.5) | 103.3 (19.6)

6. Secondary Outcome: Macrophage-derived Chemokine
Description: ELISA assay macrophage-derived chemokine
Time Frame: 6 hours
Population: plasma levels
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Cangrelor | No Cangrelor
Number analyzed (Participants) | 13 | 9
pg/mL | 593.3 (44) | 873.8 (63.8)

ADVERSE EVENTS:
Time Frame: 48 hours
Description: bleeding
Arm/Group | Cangrelor | No Cangrelor
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 0/13 | 0/9

LIMITATIONS AND CAVEATS:
The study was terminated because of slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT03043274/Prot_SAP_000.pdf